CLINICAL TRIAL: NCT00438633
Title: Early vs Delayed Physical Therapy (Exercises) for Non-Operatively-Treated Proximal Humerus Fractures: A Prospective Randomized Trial
Brief Title: Comparison of Early and Late Therapy for Adults With Non-Operatively Treated Proximal Humerus Fractures
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Neal Chung-Jen Chen, Principal Investigator; Hand Service, Massachusetts General Hospital
Other Study IDs: 2004-P-002235
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Results first posted 2019-06-21 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Proximal Humeral Fractures
Keywords: proximal humerus fracture; rehabilitation; non-operative treatment; DASH and Constant instruments
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Early Therapy: Subjects who begin therapy immediately after diagnosis of injury.
- Late Therapy: Subjects who delay therapy for 3 weeks after diagnosis of injury.

SUMMARY:
The purpose of the study is to compare two common ways of rehabilitating after proximal humerus fractures treated non-operatively.

DETAILED DESCRIPTION:
Proximal humerus fractures with limited displacement and fractures that occur in older, less active or infirm patients are treated non-operatively. There is a general impression, supported by some data, that better function is obtained with immediate initiation of shoulder exercises. However, there is some concern that this may contribute to nonunion of the fracture and may be unnecessary. Some researchers have demonstrated better outcomes with immediate rehabilitation with pendulum movements. Others have shown similar functional outcomes when rehabilitation begins approximately a month after injury, or when radiographs show signs of bone healing, and this delay is associated with lower rates of non-union and malunion occurrence.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female patients.
* Any race
* Older than 18y
* Diagnosed with proximal humeral fracture clinically and confirmed by imaging studies: X rays and/or CT Scans.
* Any type of proximal humeral fracture according to the Neer or AO classification system.
* Patient should have received non-operative treatment.

Exclusion Criteria:

* Patients younger than 18 y.
* Patients with multiple other fractures.
* Patients that have received surgical treatment including closed reduction and percutaneous fixation, open reduction and internal fixation (plates, screws, pins, tension wire bands, cerclage wiring and/or intramedullary nailing) and/or articular shoulder prosthesis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the MGH Hand and Upper Extremity or Trauma service
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2005-02 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Chen, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Early Therapy | Late Therapy
Started | 32 | 31
3-month Follow-up | 26 | 24
Completed | 16 | 14
Not Completed | 16 | 17
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 15 | 17

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are assessed for all subjects completing 3-month follow-up.
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Therapy | Late Therapy | Total
Number analyzed (Participants) | 26 | 24 | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63 (13) | 62 (12) | 63 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 21 | 15 | 36
Injured Hand [Count of Participants; unit: Participants]
  Dominant | 9 | 12 | 21
  Non-dominant | 17 | 12 | 29
Non- or minimally displaced [Count of Participants; unit: Participants]
  Yes | 22 | 19 | 41
  No | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Shoulder Flexion
Description: We measured active forward flexion of the shoulder
Time Frame: 6 months
Population: All analysis conducted with those who completed 3-month follow-up. We used mean imputation for the 6-month evaluation for patients who did not attend a 6-month follow-up.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Early Therapy | Late Therapy
Number analyzed (Participants) | 26 | 24
Degrees | 150 (26) | 146 (22)

2. Secondary Outcome: Shoulder Pain Likert Scores
Description: Rated on a scale of 0-10, where 0 is no pain and 10 is severe pain.
Time Frame: 3 months, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Early Therapy | Late Therapy
Number analyzed (Participants) | 26 | 24
units on a scale
  NRS Pain, 3 months | 3 (2) | 3 (1)
  NRS Pain, 6 months | 2 (1) | 2 (3)

3. Secondary Outcome: External Rotation
Time Frame: 3 months, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Early Therapy | Late Therapy
Number analyzed (Participants) | 26 | 24
Degrees
  External Rotation, 3 months | 53 (30) | 51 (21)
  External Rotation, 6 months | 70 (17) | 66 (26)

4. Secondary Outcome: Abduction
Time Frame: 3 months, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Early Therapy | Late Therapy
Number analyzed (Participants) | 26 | 24
Degrees
  Abduction, 3 months | 115 (43) | 101 (41)
  Abduction, 6 months | 147 (27) | 136 (33)

5. Secondary Outcome: Disability of the Hand, Shoulder, and Arm Score
Description: Disability of the Hand, Shoulder, and Arm Score (DASH) is a measure of upper extremity physical function, with scores ranging from 0 to 100. A higher score indicates more physical impairment.
Time Frame: 3 months, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Early Therapy | Late Therapy
Number analyzed (Participants) | 26 | 24
Units on a scale
  DASH, 3 months | 33 (25) | 24 (15)
  DASH, 6 months | 18 (12) | 14 (7)

ADVERSE EVENTS:
Arm/Group | Early Therapy | Late Therapy
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24
Other Adverse Events (participants affected / at risk) | 0/26 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes